CLINICAL TRIAL: NCT02966977
Title: Clinical Study To Analyse The Influence Of An Extended Urine Analysis By Mass Spectrometry On Internal Medicine Wards At The University Hospital Of Basel
Brief Title: Extending Urine Analysis By Direct Mass Spectrometry
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 2016-01534
Record Dates: First submitted 2016-11-15; First posted 2016-11-17 (Estimated); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: Urinary Tract Infection (Diagnosis)
MeSH Terms: conditions — Urinary Tract Infections; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional microbiological diagnostics (Active Comparator): Conventional microbiological identification by culture plate (overnight cultures with subsequent bacterial/fungal identification).
  Interventions: Other: Conventional microbiological identification by culture plate
- Conventional plus mass spectrometry (Experimental): Conventional microbiological identification by culture plate plus Direct mass spectrometry identification from urine sample. This additional diagnostic procedure is supplied additionally to conventional diagnostics.
  Interventions: Other: Conventional microbiological identification by culture plate; Other: Direct mass spectrometry identification from urine sample

INTERVENTIONS:
Other: Conventional microbiological identification by culture plate — Conventional microbiological identification involves a step of overnight-2days growth of bacteria/fungi on culture plates prior to identification by biochemical methods or by mass spectrometry. See also information noted in arm/group description.
Other: Direct mass spectrometry identification from urine sample — The urine sample is concentrated and directly measured by a MALDI-TOF mass spectrometer without an intermediary microbiological culture on agar plates.
  Arms: Conventional plus mass spectrometry

SUMMARY:
The aim of this study is to evaluate the effect of an extension of conventional urine diagnostics with mass spectrometry in patients with a suspected UTI. Mass spectrometry is done directly from the urine sample (without an intermediate bacterial culture).The primary outcome is the time from the entry of a urine sample in the microbiological laboratory to the adequate/optimal/definitive treatment. Secondary outcomes are the time to diagnosis of a therapy relevant UTI, the quantity of antibiotics prescribed per patient and ward and a comparison of the length of hospital stay.

DETAILED DESCRIPTION:
Urinary tract infections (UTI) have a high incidence rate and are one of the main reasons for initiating an antibiotic therapy, both, in the ambulatory and hospital setting. Mass spectrometry and improved sample preparation allows same-day identification of the causing agent of an UTI. This could shorten the time of suboptimal and potentially harmful empirical therapy. Additionally adverse effects from and the development of resistance against the applied antibiotic agent could be diminished. Matrix Assisted Laser Desorption Ionization (MALDI)- Time of Flight (TOF) Mass Spectrometry (MS) (MALDI-TOF MS) is already the preferred identification method in an increasing number of laboratories since it outperforms biochemical identification by speed and precision. This study tries to evaluate this new method to identify the causing agent of an UTI and evaluates its clinical implications.

This research project is a clinical trial that intends to analyse urine of patients with suspected urinary tract infections by mass spectrometry. This patient material is conventionally processed and not retrieved particularly for study purposes. Health-related personal data is collected from patients on the wards of the Clinic for Internal Medicine at the University Hospital Basel that have a urine sample analysed during the study period. No health-related personal data is particularly collected for this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients of the Clinic for Internal Medicine at the University Hospital Basel with a suspected UTI and a minimum of one urine sample sent to the clinical microbiology laboratory.

Additionally at least one of the following:

* Patients consented to the general (i.e. "hospital-wide") use of their data and samples for research purposes.
* Patients consented to be enrolled in this study (by being informed about this study and signing the study specific consent form).
* Patients who are exempted from the need for a consent by way of an exception in agreement to the decisions of the competent ethics committee.

Exclusion Criteria:

* Minors or persons who declined the general use of their data and samples for research purposes (hospital wide consent) and declined or did not decide on the study specific consent form are not included.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2016-10-03 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2017-04-15 (Actual)

PRIMARY OUTCOMES:
Time from the entry of a urine sample in the microbiological laboratory to the adequate/optimal/definitive treatment. | 1 week

SECONDARY OUTCOMES:
Time to diagnosis of a therapy relevant UTI. | 1 week
Quantity of antibiotics prescribed per patient and ward. | 2 weeks
Comparison of the length of hospital stay | 2 weeks
Comparison of the number of possible complications connected to UTI | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Egli, PD Dr. FAMH, Principal Investigator — Clinical Microbiology, University Hospital Basel
Locations (1):
- University Hospital Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No